CLINICAL TRIAL: NCT03224364
Title: A Randomized Controlled Trial Comparing a Solo and Non-solo Approach for Laparoscopic Appendectomy
Brief Title: Solo and Non-solo Approach for Laparoscopic Appendectomy (SOLOAP)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Say-June Kim (Other)
Responsible Party: Sponsor-Investigator, Say-June Kim, Professor, Daejeon St. Mary's hospital
Organization: Daejeon St. Mary's hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SSAP-1
Record Dates: First submitted 2017-07-18; First posted 2017-07-21 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Appendicitis; Laparoscopic
Keywords: Solo surgery; Camera holder; Laparoscopic Appendectomy
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LC & nonsolo approach (Placebo Comparator): The surgical intervention is nonsolo LC
  Interventions: Procedure: nonsolo LA
- LC & solo approach (Active Comparator): The surgical intervention is solo LC.
  Interventions: Procedure: solo LA

INTERVENTIONS:
Procedure: nonsolo LA — This patient is scheduled to undergo nonsolo laparoscpic appendectomy.
  Other Names: Nonsolo laparoscopic appendectomy
  Arms: LC & nonsolo approach
Procedure: solo LA — This patient is scheduled to undergo solo laparoscpic appendectomy.
  Other Names: Solo laparoscopic appendectomy
  Arms: LC & solo approach

SUMMARY:
To determine the safety and feasibility of solo laparoscopic appendectomy, which is defined as the application of solo surgery to laparoscopic appendectomy, by comparing consecutive non-solo procedures conducted by a surgeon in the presence or absence of human assistant(s).

DETAILED DESCRIPTION:
Laporoscopic appendectomy usually requires three surgeons, including an operator, a camera assistant, and other instrument assistant. Recent advancement of technology made it possible to develop the conveniently adjustable holders for camera and other laparoscopic instruments. The application of these instruments enables "solo-surgery" wherein an operation is driven by single surgeon. During surgery, human assistant(s) are helpful because of their instant assistance according to the operation's need. Therefore, the utilization of instruments instead of human assistants would be cumbersome. However, the utilization of instruments would be helpful by enabling operation-driven repositioning of the camera and instrument(s). Currently, no attempt has been made to objectively compare the merits and demerits of these two procedures. Therefore, this study was conducted to determine the safety and feasibility of solo laparoscopic appendectomy, which is defined as the application of solo surgery to laparoscopic appendectomy, by comparing consecutive non-solo procedures conducted by a surgeon in the presence or absence of human assistant(s).

ELIGIBILITY:
Inclusion Criteria:

1. The patients planned to undergo elective laparoscopic appendectomy
2. Benign gallbladder diseases requiring surgery
3. The patients who are indicated for single-port laparoscopic appendectomy.

Exclusion Criteria:

1. the patients with complicated cholecystitis
2. the patients with the gallbladder with a thickness more than 4mm.
3. the patients who are expected to have severe peritoneal adhesion.
4. the patients with malignant gallbladder diseases.
5. the patients whose operation appears to need human assistant(s)

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2017-08-01 (Estimated); Primary Completion 2017-12-31 (Estimated); Study Completion 2018-03-31 (Estimated)

PRIMARY OUTCOMES:
Operation time | day 1
  Operation time correlates with surgical difficulity.

SECONDARY OUTCOMES:
Pain score | day 3
  Daily pain scores are assessed

CONTACTS AND LOCATIONS:
Overall Officials: Say-June Kim, M.D., Ph.D., Principal Investigator — Daejeon St. Mary's hospital, the Catholic University of Korea, 222, Banpo-dong, Seocho-gu, Seoul, 06591, South Korea

IPD SHARING:
Plan to Share IPD: No